CLINICAL TRIAL: NCT04292041
Title: Fasting Mimicking Diet in Prostate Cancer and Metabolic Syndrome, a Pilot Study
Brief Title: Fasting Mimicking Diet in Prostate Cancer and Metabolic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Galway Clinic (Network)
Responsible Party: Principal Investigator, Professor Frank Sullivan, Medical Director, Department of Radiation Oncology, Galway Clinic
Other Study IDs: GalwayC
Record Dates: First submitted 2020-02-21; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Prostate Cancer; Metabolic Syndrome; Intermittent Fasting
Keywords: Fasting Mimicking Diet
MeSH Terms: conditions — Prostatic Neoplasms; Metabolic Syndrome; Intermittent Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fasting mimicking diet — 3 cycles of programmed nutrition using a fasting mimicking diet (Chemolieve (R)), each cycle consisting of 4 days. Pre and post nutritional cycles, clinical and metabolic assessments are taken, as per protocol. Allowing for a 3 month "washout" time, the 'post' assessment is planned approximately 6 months from the initial (pre) assessment.
  Other Names: Programmed cyclic nutrition for 3 monthly cycles (fasting mimicking diet)

SUMMARY:
This is a prospective observational cohort study of patients with prostate cancer who have a metabolic syndrome. The study aims to evaluate the role of intermittent fasting (fasting mimicking diet) in these patients. The primary end point is metabolic health and the secondary endpoint is quality of life.

DETAILED DESCRIPTION:
Cancer is a complex set of conditions which collectively comprise the second biggest cause of death in the western world. In addition, these diseases, along with their various treatments, are associated with significant illness, as well as a host of debilitating symptoms. Two very common problems are cancer fatigue, as well as metabolic changes which can cause much suffering in and of themselves. Patients with advanced cancers, as well as many patients undergoing surgery, radiation therapy as well as chemotherapy all complain of fatigue, to a greater or lesser extent. Many gain or lose weight, and develop associated metabolic changes in uninvolved body systems, which can cause a significant health burden on the patients, as well as the healthcare system as a whole.

Little is known about the mechanisms which underlie these symptoms. Various biologic processes have been implicated including inflammation and other changes in body metabolism. There is urgent need to better understand these processes, which cause so much suffering in cancer patients, so as to potentially develop more effective solutions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven prostate cancer having features of a metabolic syndrome, receiving standard treatment options for their disease.

Exclusion Criteria:

* Patients without a diagnosis of prostate cancer
* Life expectancy less than 1 year
* Children under the age of 18
* Individuals who are allergic to nuts or soy
* Individuals with a Body Mass Index (BMI) <18.5
* Individuals who have been severely weakened by a disease or medical procedure
* Individuals who are taking medications which may not be safely consumed with a calorie restricted diet unless authorised in writing by a licensed physician
* Individuals with a history of significant cardiac disease, particularly uncompensated congestive heart failure NYHA grade 2 or more or LVEF <40% on any prior assessment
* Individuals with a history of syncope (fainting) with calorie restriction or other medical co-morbidities
* Individuals who have special dietary needs that are incompatible with the ProLon® meal plan
* Individuals with liver or kidney disorders that may be affected by the very low glucose and protein content of the diet

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: A cohort of 40 men with biopsy-proven prostate cancer having features of a metabolic syndrome, receiving standard treatment options for their disease.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in Baseline Weight (in kilograms) at 6 months | Baseline and 3 months after Nutritional Cycle 3 (each cycle is 4 days per month), about 6 months
  Metabolic health parameter
Change in Baseline Blood Pressure (in millimeters of Mercury) at 6 months | Baseline and 3 months after Nutritional Cycle 3 (each cycle is 4 days per month), about 6 months
  Metabolic health parameter
Change in Baseline Waist Circumference (in centimeters) at 6 months | Baseline and 3 months after Nutritional Cycle 3 (each cycle is 4 days per month), about 6 months
  Metabolic health parameter
Change in Baseline Triglycerides Level (in millimoles per litre) at 6 months | Baseline and 3 months after Nutritional Cycle 3 (each cycle is 4 days per month), about 6 months
  Clinical lab results
Change in Baseline Total, LDL, and HDL Cholesterol (in millimoles per litre) at 6 months | Baseline and 3 months after Nutritional Cycle 3 (each cycle is 4 days per month), about 6 months
  Clinical lab results

SECONDARY OUTCOMES:
Change in Baseline EQ5D5L Health Questionnaire Score at 6 months | Baseline and 3 months after Nutritional Cycle 3 (each cycle is 4 days per month), about 6 months
  Structured Quality of Life Measure - Patients' self report of mobility, self-care, usual activities, pain/discomfort, anxiety/depression -
  1. No problem
  2. Slight problems
  3. Moderate problems
  4. Severe problems
  5. Unable to/extreme problems
     * 5 questions
     * Minimum score of 0, meaning good quality of life
     * Maximum score of 25, meaning poor quality of life
Change in Baseline EQ5D5L Vertical Visual Analogue Scale Score at 6 months | Baseline and 3 months after Nutritional Cycle 3 (each cycle is 4 days per month), about 6 months
  Structured Quality of Life Measure - Patients' self report on how good/bad their health is TODAY -
  * One scale numbered from 0 to 100
  * Minimum score of 0, meaning the worst health you can imagine
  * Maximum score of 100, meaning the best health you can imagine
Change in Baseline Chalder Fatigue Index Score at 6 months | Baseline and 3 months after Nutritional Cycle 3 (each cycle is 4 days per month), about 6 months
  Structured Tiredness/Fatigue Measures on Likert Scale - Patients' self report of fatigue symptoms -
  0: Less than usual
  1. No more than usual
  2. More than usual
  3. Much more than usual
     * 6 questions
     * minimum score of 0, meaning no fatigue due to illness
     * maximum score of 18, meaning chronic fatigue due to illness

CONTACTS AND LOCATIONS:
Overall Officials: Frank Sullivan, MSc, Principal Investigator — Galway Clinic
Locations (1):
- Galway Clinic, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No
None planned

REFERENCES:
- [Result] Brandhorst S, Longo VD. Protein Quantity and Source, Fasting-Mimicking Diets, and Longevity. Adv Nutr. 2019 Nov 1;10(Suppl_4):S340-S350. doi: 10.1093/advances/nmz079. PMID 31728501
- [Result] Fontana L, Partridge L, Longo VD. Extending healthy life span--from yeast to humans. Science. 2010 Apr 16;328(5976):321-6. doi: 10.1126/science.1172539. PMID 20395504
- [Result] Mirzaei H, Suarez JA, Longo VD. Protein and amino acid restriction, aging and disease: from yeast to humans. Trends Endocrinol Metab. 2014 Nov;25(11):558-66. doi: 10.1016/j.tem.2014.07.002. Epub 2014 Aug 19. PMID 25153840
- [Derived] Fay-Watt V, O'Connor S, Roshan D, Romeo AC, Longo VD, Sullivan FJ. The impact of a fasting mimicking diet on the metabolic health of a prospective cohort of patients with prostate cancer: a pilot implementation study. Prostate Cancer Prostatic Dis. 2023 Jun;26(2):317-322. doi: 10.1038/s41391-022-00528-3. Epub 2022 Mar 21. PMID 35314788